CLINICAL TRIAL: NCT05597930
Title: Development and Validation of a New Wrist Orthosis by 3D Printing
Brief Title: New 3D Printed Wrist Orthosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: TOPMED (Other)
Collaborators: Medicus (Unknown); Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RD-21-0376
Record Dates: First submitted 2022-10-20; First posted 2022-10-28 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Carpal Tunnel Syndrome; Ulnar Nerve Injury; Rhizarthrosis; Tendinopathy, Thumb; Tenosynovitis de Quervain; Hand Disease
MeSH Terms: conditions — Carpal Tunnel Syndrome; Tendinopathy; De Quervain Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thumb then wrist orthosis (Experimental)
  Interventions: Device: Wrist and Thumb orthosis
- Wrist then thumb orthosis (Experimental)
  Interventions: Device: Wrist and Thumb orthosis

INTERVENTIONS:
Device: Wrist and Thumb orthosis — Custom 3D printed thumb and wrist orthosis

SUMMARY:
In order to offer a new product improving the healing and/or rehabilitation of injuries or injuries to the wrist and hand, Médicus is seeking to develop a new orthosis for the wrist and hand by 3D printing. This project will focus on the development of an orthosis related to carpal tunnel syndrome as well as droopy hand. Among the issues to be addressed in this development proposal, the investigators find: 1) Identification of the best methodology for taking digital impressions; design of an orthosis with the following characteristics: (i) no external attachment system, (ii) spiral design with a thumb ring, (iii) manufacturing by 3D printing and (iv) a cost of less than $150 ;3) Performing technical and clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 70 years old
* Ability to accurately communicate comfort and discomfort,
* Carpal tunnel syndrome, or
* de Quervain's tenosynovitis, or
* Drop hand, or
* Ulnar nerve damage
* Rhizarthrosis, or
* Tendinopathy of the thumb
* And/or ulnar gale

Exclusion Criteria:

* - Spasticity in the upper limbs
* Paralysis, Insensitivity of the upper limbs
* Neuromuscular pathology affecting the upper limbs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2024-05-24 (Estimated); Study Completion 2024-05-24 (Estimated)

PRIMARY OUTCOMES:
Change in pain during treatment from baseline at day 14 | Baseline and day 14
  Pain measure via 1-5 rating, possible scores range from1 (no pain) to 5 (worst possible pain). Change = (Day 14 score - baseline score)

SECONDARY OUTCOMES:
Difficulty in donning the orthosis | Each day during 2 weeks of intervention
  Yes/No question about having difficulty putting on the orthosis. No unit.
Comfort | Each day during 2 weeks of intervention
  Comfort measure via 1-5 rating, possible scores range from1 (worst possible comfort) to 5 (best possible comfort). No unit.
Weight satisfaction rating at baseline | Baseline
  Weight satisfaction measure via 1-5 rating, possible scores range from1 (worst possible satisfaction) to 5 (best possible satisfaction). No unit.
Satisfaction on ease of donning | Baseline
  Satisfaction measure via 1-5 rating on ease of donning, possible scores range from 1 (worst possible satisfaction) to 5 (best possible satisfaction). No unit.
Satisfaction on ease of donning | Day 14 of intervention
  Satisfaction measure via 1-5 rating on ease of donning, possible scores range from 1 (worst possible satisfaction) to 5 (best possible satisfaction). No unit.
Satisfaction on ease of doffing | Baseline
  Satisfaction measure via 1-5 rating on ease of doffing, possible scores range from 1 (worst possible satisfaction) to 5 (best possible satisfaction). No unit.
Satisfaction on ease of doffing | Day 14 of intervention
  Satisfaction measure via 1-5 rating on ease of doffing, possible scores range from 1 (worst possible satisfaction) to 5 (best possible satisfaction). No unit.
Functional disability evaluation of the upper member | Baseline
  Evaluation of disability of arm, shoulder and hand in activities of daily living via Quick Disability of arm, shoulder and hand (Quick DASH) (validated 11 elements 5-point rating). Possible scores range from 1 (No difficulty) to 5 (Incapacity to complete task). No unit.
Functional disability evaluation of the upper member | Day 14 of intervention
  Evaluation of disability of arm, shoulder and hand in activities of daily living via Quick Disability of arm, shoulder and hand (Quick DASH) (validated 11 elements 5-point rating). Possible scores range from 1 (No difficulty) to 5 (Incapacity to complete task). No unit.
Weight satisfaction rating at day 14 of intervention | Day 14 of intervention
  Weight satisfaction measure via 1-5 rating, possible scores range from1 (worst possible satisfaction) to 5 (best possible satisfaction). No unit.
aesthetic satisfaction rating at day 14 of intervention | Day 14 of intervention
  Aesthetic satisfaction measure via 1-5 rating, possible scores range from1 (worst possible satisfaction) to 5 (best possible satisfaction). No unit.
aesthetic satisfaction rating at baseline | Baseline
  Aesthetic satisfaction measure via 1-5 rating, possible scores range from1 (worst possible satisfaction) to 5 (best possible satisfaction). No unit.
material quality satisfaction rating at baseline | Baseline
  Material quality satisfaction measure via 1-5 rating, possible scores range from1 (worst possible satisfaction) to 5 (best possible satisfaction). No unit.
material quality satisfaction rating at day 14 of intervention | Day 14 of intervention
  Material quality satisfaction measure via 1-5 rating, possible scores range from1 (worst possible satisfaction) to 5 (best possible satisfaction). No unit.

CONTACTS AND LOCATIONS:
Locations (1):
- TOPMED, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No